CLINICAL TRIAL: NCT01624701
Title: Clinical Ex Vivo Expansion of Human Umbilical Cord Blood Stem and Progenitor Cells: A Pilot Trial in Collaboration With the Massachusetts Institute of Technology
Brief Title: Clinical Ex Vivo Expansion of Human Umbilical Cord Blood Stem and Progenitor Cells
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding expired
Sponsor: Singapore General Hospital (Other)
Collaborators: Whitehead Institute for Biomedical Research (Unknown); Blood Services Group, Health Sciences Authority of Singapore (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009/925/B
Record Dates: First submitted 2012-03-20; First posted 2012-06-21 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Acute Leukemia; Chronic Leukemia; Myelodysplastic Syndrome; Lymphoma; Myeloma
Keywords: Cord blood; unrelated donor; allogeneic; cell dose
MeSH Terms: conditions — Myelodysplastic Syndromes; Lymphoma; Neoplasms, Plasma Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Expanded (Experimental): 'Ex vivo expanded cord blood cells
  Interventions: Other: Ex vivo expanded cord blood cells

INTERVENTIONS:
Other: Ex vivo expanded cord blood cells — Cord blood cells will be expanded ex vivo using a combination of stem cell factor (SCF), thrombopoietin (TPO), Flt3 ligand and IGFBP2 with mesenchymal stromal cell (MSC) co-culture.

SUMMARY:
This is a pilot clinical trial to assess the feasibility and efficacy of expanding umbilical cord blood derived blood stem cells for transplantation using a combination of chemical factors and stromal co-culture. Bone marrow (BM) mesenchymal stromal cells (MSC) will be obtained from a separate bone marrow donor. One cord blood unit will be expanded by this method while another cord blood unit will be infused without manipulation. The expanded cord blood unit will help boost the initial recovery of blood counts after transplantation, though it is expected that the unexpanded cord blood unit will provide the cells which will lead to long term engraftment of blood stem cells. A third cord blood unit will be identified for standby should the cord blood unit expansion fail.

DETAILED DESCRIPTION:
1. Clinical transplantation of two cord blood units: one ex vivo expanded while another unmanipulated unit to function as a back-up.
2. Ten patients will be selected from those for whom:

   * Allogeneic haematopoietic stem cell transplant is indicated (see details)
   * No matched sibling or matched unrelated donor is available quickly enough for the transplant (no fully matched donor found within 1 month of initiation of donor search or donor found but not available for donation within 3 months of donor search).
   * At least three unrelated donor cord blood unit can be identified with less than 2 antigens mismatches with the patient but with insufficient cell dose to meet the patient's requirements. If clinical efficacy of this protocol is demonstrated, we will proceed to a multicentre clinical trial with more patients.
3. The investigators will obtain haplo-identical MSC from the bone marrow of sibling/parent/offspring of the patient. Although there will be some MSC co-infused with the cord blood cells, this has been shown to be safe in trials of MSC given for patients with graft versus host disease (GVHD) and human leukocyte antigen (HLA) matching of MSC and recipient has been shown to be not important. bone marrow mesenchymal stroma cells (BM-MSCs) derived from related donor bone marrow with a minimum of 2/6 HLA match have been safe for use in patients.1 If the haplo-identical MSC donor is not available, matched unrelated donor MSC would also be used.
4. Efficacy will be assessed by the following and compared to published literature as well as historical controls:

   * Neutrophil and platelet engraftment
   * Post transplant 100-day mortality
   * Overall and progression-free survival If clinical efficacy of this protocol is demonstrated, the investigators will proceed to a multicentre clinical trial with more patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be from the Department of Haematology, Singapore General Hospital, who have the diagnoses listed below and who meet the inclusion criteria. They have to be deemed suitable for trial by the respective attending doctor as well as a panel of at least three hematologists. Suitability will be reassessed by the Principal Investigator again

  1. Patients aged 12 years to 60 years.
  2. Patient has no currently available HLA-A, B, C, DRB1 and DQB1 matched related or unrelated donor.
  3. Patient must have a hematologic malignancy requiring allogeneic haematopoietic stem cell transplantation as further defined below (from National Marrow Donor Program and American Society of Blood and Marrow Transplantation Guidelines) and as further agreed upon by a panel of at least three hematologists specializing in transplantation.
* Acute myelogenous leukemia (AML): High-risk AML including:

  * Antecedent hematological disease (e.g., myelodysplasia (MDS))
  * Treatment-related leukemia
  * Induction failure
  * 1st complete remission (CR1) with poor-risk cytogenetics or molecular markers (e.g. Flt 3 mutation, 11q23 etc)
  * 2nd complete remission (CR2) and beyond
* Acute lymphoblastic leukemia (ALL)

  * CR1 up to age 35
  * High-risk over age 35 including:
  * Poor-risk cytogenetics (e.g., Philadelphia chromosome t(9;22)or 11q23 rearrangements)
  * High white cell count (> 30,000/mm3) at diagnosis
  * CNS or testicular leukemia
  * No CR within 4 weeks of initial treatment
  * Induction failure
  * CR2 and beyond
* Myelodysplastic syndromes (MDS)

  * Intermediate-1 (INT-1), intermediate-2 (INT-2) or high IPSS score which includes:
  * > 5% marrow blasts
  * Other than good risk cytogenetics (not 5q- or normal)
  * > 1 lineage cytopenia
* Chronic myelogenous leukemia (CML)

  * Disease progression
  * Accelerated phase
  * Blast crisis (myeloid or lymphoid)
* Follicular lymphoma

  * Poor response to initial treatment
  * After second or subsequent relapse
  * Transformation to diffuse large B-cell lymphoma
* Aggressive T-cell or B-Cell lymphoma

  * After second or subsequent relapse
  * No CR with initial treatment
* Mantle Cell: After second or subsequent relapse
* Hodgkin's lymphoma

  * No initial CR
  * After second or subsequent relapse
* Multiple myeloma: Patients failing autologous transplantation with chromosome 13 abnormalities, first response lasting less than 6 months, or β-2 microglobulin > 3 mg/L may be considered for this protocol after initial therapy.

Exclusion Criteria:

1. Inadequate Organ Function as defined by:

   * Renal: Creatinine clearance > 60ml/min
   * Hepatic: Bilirubin, AST/ALT < 2x upper limit of normal
   * Pulmonary function: DLCOcorr > 50% normal
   * Cardiac: left ventricular ejection fraction > 45%
2. Karnofsky score (adults) < 70% or Lansky score < 50% (pediatrics)

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2012-03; Primary Completion 2015-07 (Actual); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Safety | 1 month
  Number of subjects with infusional toxicities (including fever, renal dysfunction within 72 hours of infusion) and potential immunologic competition (absent chimerism of donor cells by 21 days post transplantation).

SECONDARY OUTCOMES:
Engraftment | 2 months
  Neutrophil engraftment (ANC>500/ul) in subjects as demonstrated by number of subjects with engraftment <=21 days.

CONTACTS AND LOCATIONS:
Overall Officials: William YK Hwang, MBBS, FRCP, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore